CLINICAL TRIAL: NCT05610566
Title: A Prospective, Multicentric Clinical Trial Protocol to Evaluate the Safety and Efficacy of the HighLife Trans-Septal Transcatheter Mitral Valve Replacement System for the Treatment of Moderate-severe or Severe Mitral Regurgitation With Single-arm Objective Performance Criteria
Brief Title: Safety and Efficacy of the HighLife Transcatherter Mitral Valve Replacement System in Patients With Moderate-severe or Severe Mitral Regurgitation in China
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peijia Medical Technology (Suzhou) Co., Ltd. (Industry)
Collaborators: West China Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); The Second Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23CSP001
Record Dates: First submitted 2022-11-01; First posted 2022-11-09 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A single set of test (Experimental): The HighLife Trans-Septal TMVR System comprises a 28mm Transcatheter Mitral Valve, a loop placement catheter, a sub-annular implant and its delivery systems.
  Interventions: Device: the HighLife Trans-Septal Transcatheter Mitral Valve Replacement System

INTERVENTIONS:
Device: the HighLife Trans-Septal Transcatheter Mitral Valve Replacement System — The HighLife TMVR system is composed of a Transcatheter Mitral Valve (TMV), a subannular implant (SAI), and their delivery systems and accessories. The TMV is a 28mm mitral bioprosthesis made of a self-expanding Nitinol frame covered with polyester graft and supporting bovine pericardium leaflets. The bioprosthesis is used in conjunction with the Sub-Annular Implant (SAI), comprising a ring (made of polycarbonate urethane (PCU), nitinol, gold markers and polyester (Dacron) to be placed around the mitral valve apparatus to stabilize the position of the mitral valve implant.

SUMMARY:
To observe and evaluate the safety and efficacy of the HighLife Transcatheter Mitral Valve Replacement System in patients with moderate-severe or severe mitral valve regurgitation through a prospective, multicenter clinical trial using objective performance criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who voluntarily participate and sign the informed consent form and can cooperate with the completion of the entire trial process;
2. Age ≥ 18 years old;
3. Moderate-severe or severe mitral regurgitation (≥3+); Note 1: Patients with ischemic or non-ischemic heart disease induced symptomatic secondary mitral regurgitation as the primary cause must be treated for at least 1 month after optimal guideline medical therapy (GDMT). Echocardiography should be performed 3 months after cardiac resynchronization therapy and 1 month after coronary revascularization to assess the degree of regurgitation.

   Note 2: For patients with primary mitral regurgitation, the multidisciplinary cardiac team of the research center needs to use a standard scoring system, considering multiple factors such as complications, frailty, and disability, ensuring the enrolled with a high risk of surgery.
4. Patients with New York Heart Association (NYHA) functional ratings are Class II, III, or ambulatory Class IV;
5. Anatomically appropriate for treatment with the HighLife Transcatheter Mitral Valve Replacement System.

Exclusion Criteria:

1. Patients had any stroke/TIA within 30 days;
2. Patients with severe symptomatic bilateral carotid stenosis (>70% stenosis on non-invasive imaging);
3. Patients with active infection requiring antibiotic therapy;
4. Patients with active ulcer or gastrointestinal bleeding within the past 3 months;
5. Patients with history of coagulopathy or refuse future blood transfusion;
6. Patients unable to undergo transesophageal echocardiography (TEE);
7. Patients who are pregnant or breastfeeding, or planning to have children within 12 months;
8. Patients who are unable to adhere to the follow-up schedule and complete the examination;
9. Patients enrolled in other clinical studies and within the follow-up period;
10. Patients with known allergies to device components or contrast agents;
11. Patients unable to receive anticoagulant or antiplatelet therapy;
12. Patients with a life expectancy of less than 12 months due to non-cardiac disease;
13. Patients requiring emergency surgical treatment;
14. Patients scheduled for cardiac surgery within 12 months;
15. Patients with an inappropriate mitral annulus or leaflet size (<30 mm and >45 mm);
16. Patients with moderate or above mitral stenosis;
17. Flail mitral leaflets, or moderate to severe mitral valve prolapse;
18. Patients with severe hepatic or renal insufficiency;
19. Patients with severe calcification of the mitral annulus and/or mitral leaflets;
20. Patients with history of mitral valve surgery or interventional therapy, or left atrial appendage occlusion device;
21. Patients had acute myocardial infarction (MI) (Q-wave MI, or non-Q-wave MI, with CK-MB twice the normal and/or T-MB) within the past 1 month;
22. Patients with untreated symptomatic coronary lesions requiring revascularization;
23. Patients with untreated severe aortic stenosis and severe aortic regurgitation;
24. Patients with aortic valve prosthesis;
25. Patients with severe tricuspid valve lesions requiring surgical intervention;
26. Patients with significant right ventricular dysfunction (such as biliteral lower extremities edema with increased jugular vein pulsation and hepatomegaly;
27. LVEF < 30%; LVEDD > 70 mm;
28. Patients with echocardiographically confirmed intracardiac mass, thrombus or neoplasm;
29. Hypertrophic obstructive cardiomyopathy (HOCM);
30. Patients with active or recent (within 3 months) endocarditis;
31. Patients with definite non-left heart disease induced severe pulmonary hypertension (echocardiographic indication: systolic pulmonary artery pressure (SPAP) > 70 mmHg)
32. Patients with hypotension (systolic blood pressure <90 mmHg) occurring within 7 days or mechanical hemodynamic support.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2025-07-06 (Estimated); Study Completion 2029-07-06 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality at 12 months | 12 months
  All-cause mortality

SECONDARY OUTCOMES:
Technical success | Immediate after procedure
  Technical success defined as an alive patient at exit from procedure room, with all of the following:
  * Successful vascular access, delivery and retrieval of the HighLife delivery systems
  * Deployment and correct positioning of the HighLife 28mm bioprosthesis
  * Freedom from additional emergency surgery or re-intervention related to the device or access procedure, that occurred (was initiated) during the procedure. Any emergency surgery or re-intervention that occurs after the patient exits the procedure room/cath lab in stable condition will be captured as an AE/SAE.
Cardiac function change | 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years
  NYHA functional classification
Quality of life of patients | 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years
  Quality of Life of patients accessed by EuroQol-5 Dimensions (EQ-5D) Questionnaire. The higher scores mean a worse health state. Recording changes from baseline.

OTHER OUTCOMES:
Operative complication | Immediately after procedure
  The rate of operative complication
The incidence of major adverse cardiovascular and cerebrovascular events during the trial(MACCEs) | 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years
  Incidence of MACCEs (mortality, stroke, myocardial infarction, and so on surgery, arrhythmias, conduction blocks) during the trial
Incidence of major adverse valve-related events (MAVREs) during the trial | 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years
  including prosthetic valve-related death, permanent cardiac pacemaker implantation, permanent cardiac defibrillator implantation, prosthetic valve embolism, prosthetic valve thrombosis, prosthetic valve dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Peiga Medical Technology (Suzhou) Co., Suzhou, Jiangsu, China